CLINICAL TRIAL: NCT01040039
Title: Pilot Study to Assess Gut Mucosal B Cells in Individuals Co-Infected With HCV and HIV
Brief Title: Pilot Study to Assess Gut Mucosal B Cells in Individuals With HCV and HIV
Status: Terminated | Type: Observational
Why Stopped: Investigator left Rockefeller University
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: ECH-0675
Record Dates: First submitted 2009-11-19; First posted 2009-12-25 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections; Hepatitis C Virus
Keywords: HCV; HIV
MeSH Terms: conditions — HIV Infections; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, mucosal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV+HIV+
- HCV+HIV-

SUMMARY:
This pilot study aims to study gut B cells in HCV+HIV+, HCV+HIV-, HCV-HIV+, and HCV-HIV- volunteers. Volunteers will undergo a screening blood draw and flexible sigmoidoscopy with biopsy.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infects approximately 170 million people worldwide and is the leading indication of liver transplantation in the United States. HCV is primarily a blood-borne infection, and heterosexual transmission is rare. However, acute HCV infection is increasingly being reported among HIV-positive men who have sex with men (MSM) with no risk factors for parenteral HCV transmission, suggestive of a possible mucosal route of infection in these individuals. While it is possible that HCV may be transmitted into the bloodstream via mucosal tears induced by sexual activity, is also possible that a mucosal immune defect predisposes HIV+ persons to mucosal HCV transmission. Our pilot study aims to study gut B cells in HCV+HIV+, HCV+HIV-, HCV-HIV+, and HCV-HIV- volunteers. Volunteers will undergo a screening blood draw and flexible sigmoidoscopy with biopsy. We will isolate peripheral and mucosal mononuclear cells and we will perform HCV-specific ELISPOT and single B cell immunoglobulin (Ig) RT-PCR to assess volunteers' gut B cell repertoire. If successful, we would like to expand the study so as to better assess Ig repertoire differences among HCV+HIV+ and HCV+HIV- individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years of age.
2. Ability to give informed consent.
3. Platelets greater than 70,000/mm3.
4. Hb at least 9.5 g/dl.
5. INR < 1.5.

Exclusion Criteria:

1. Decompensated cirrhosis.
2. Serious uncontrolled medical illness.
3. Ingestion of Aspirin within 72 hours of sigmoidoscopy
4. Ingestion of non aspirin NSAIDS within 8 hours of sigmoidoscopy
5. Receipt of immune modulators or suppressors within 30 days prior to study entry, including, but not limited to, interferons and thalidomide.
6. Psychiatric illness or social condition that, in the opinion of the investigator, would interfere with adherence to study requirements.
7. Alcohol or drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
8. Medical illness requiring prescribed Aspirin or NSAIDs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Numbers of HCV-specific gut mucosal B cells in HCV+HIV+, compared to HCV+HIV- subjects | one year

SECONDARY OUTCOMES:
Numbers of HCV-specific gut mucosal B cells in HCV-HIV+ and HCV-HIV- subjects | 1 year
Distribution of gut mucosal B cell Ig gene segment usage in HCV+HIV+, compared to HCV+HIV- subjects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Charles, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States